CLINICAL TRIAL: NCT04522076
Title: Prospective Hospital Registry of Patients With Suspected or Confirmed Coronavirus Infection (COVID-19) and Community-acquired Pneumonia
Acronym: TARGET-VIP
Status: Active, not recruiting | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: National Medical and Surgical Center named after N.I. Pirogov of the Ministry of Healthcare of the Russian Federation (Unknown)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 02-07/20
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID-19 with pneumonia: patients with positive COVID 19 by PCR and pneumonia by CT
- COVID-19 without pneumonia: patients with positive COVID 19 by PCR and absent of pneumonia by CT
- Patients with pneumonia and without COVID 19: patients with negative COVID 19 by PCR and with pneumonia by CT
- Patients without pneumonia and COVID 19: Patients with suspected COVID-19 and/or pneumonia at the pre-hospital stage that were not confirmed in hospital

SUMMARY:
Coronavirus-2019 disease (COVID-19) and community-acquired pneumonia are significant problems of modern medicine. Pneumonia is the most common severe complication of COVID-19. But at the same time, COVID-19 is not the only cause of community-acquired pneumonia. Moreover, pneumonia is only one of the numerous possible severe complications of COVID-19. Medical centers specialized for the hospital treatment of patients with severe COVID-19 and community-acquired pneumonia were organized in different regions of Russia during coronavirus pandemic-2020. The indications for hospitalization to one of these centers based in the National Medical and Surgical Center (NMSC) are: confirmed or suspected severe COVID-19 or community-acquired pneumonia.

A prospective medical registry of such patients hospitalized to NMSC, is intended to analyze and compare their clinical and instrumental data, co-morbidity, treatment, short-term and long-term outcomes in real clinical practice.

Stage 1. Hospital treatment in NMSC

Duration of this stage: from the date of admission to the hospital up to the date of discharge from the hospital / or up to the date of death during the reference hospitalization. The date of admission to the hospital will be the date of enrollment to the study.

Evaluation of electronic health record data using the Medical Information System (MIS). Assessment of the outcomes of the hospital phase (discharge from the hospital, death) and significant events (acute respiratory and pulmonary failure, requiring mechanical ventilation; cardiovascular events - myocardial infarction, cerebral stroke, acute heart failure, paroxysmal heart rhythm disturbances, bleedings, thrombosis of large vessels and thromboembolic complications). A survey of patients to clarify data on risk factors, somatic diseases, and drug therapy before hospitalization.

COVID-19 was diagnosed when severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection was confirmed by Polymerase chain reaction (PCR). Pneumonia was confirmed according to computerized tomography (CT) data.

Stage 2. Prospective outpatient follow-up for 24 months

Duration of this stage: 24 months after discharge from the hospital This work will be delivered by investigators from the National Medical Research Center for Therapy and Preventive Medicine.

Evaluation of long-term outcomes and events among residents of Moscow and the Moscow Region according to a patient survey (contact by phone for 30-60 days, 6 months, 12 and 24 months after discharge from the hospital) and medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized to the National Medical and Surgical Center named after N.I.Pirogov of the Ministry of Health of Russia (NMSC) with suspected or confirmed COVID-19 or community-acquired pneumonia.
2. Age 18 years and older.
3. Permanent residency in Russia.

Exclusion Criteria:

1. Permanent residency outside of Russia.
2. The patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 6, 2020 until the end of the work period of departments of NMSC, that are specialized for the treatment of patients with COVID-19 and community-acquired pneumonia all patients with inclusion criteria and who don't have exclusion criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Time to all-cause mortality or Artificial Pulmonary Ventilation (APV) | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Time to all-cause mortality, nonfatal myocardial infarction, nonfatal cerebral stroke, and coronary or carotid revascularization | from discharge up to two years after reference hospitalization

SECONDARY OUTCOMES:
Proportion of patients with severe pneumonia | from admission to discharge or death during reference hospitalization, assessed up to 90 days
  Damage area >50% according to the computer tomography data at any time point during hospitalization
Proportion of patients with low oxygen saturation value | from admission to discharge or death during reference hospitalization, assessed up to 90 days
  SpO2 <90% - at any point during hospitalization
Proportion of patients with Hb <90 g/l (9.0 g/dl) at any point during hospitalization | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Proportion of patients hospitalized or transferred to Intensive Care Unit (ICU) | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Overall survival | from discharge up to two years after reference hospitalization
Time to nonfatal myocardial infarction, nonfatal cerebral stroke, and coronary or carotid revascularization | from discharge up to two years after reference hospitalization
Time to pneumonia/recurrent pneumonia | from discharge up to two years after reference hospitalization
  In patients with pneumonia during reference hospitalization time to recurrent pneumonia. In patients without pneumonia during reference hospitalization - time to first pneumonia
Time to primary or recurrent coronavirus infection disease (COVID-19) | from discharge up to two years after reference hospitalization
  In patients without COVID-19 - time to primary diagnosis and in patients with COVID-19 - time to recurrent event

OTHER OUTCOMES:
proportion of patients with nonfatal myocardial infarction | from admission to discharge or death during reference hospitalization, assessed up to 90 days
proportion of patients with nonfatal cerebral stroke | from admission to discharge or death during reference hospitalization, assessed up to 90 days
proportion of patients with bleedings | from admission to discharge or death during reference hospitalization, assessed up to 90 days
thromboembolic events | from admission to discharge or death during reference hospitalization, assessed up to 90 days
  proportion of patients with thromboembolic events
Duration of Artificial Pulmonary Ventilation | from admission to discharge or death during reference hospitalization, assessed up to 90 days
  the sum of the days when the patients required artificial pulmonary ventilation
Minimal value of oxygen blood saturation (SpO2) during the hospital stage. | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Minimal value of hemoglobin (Hb) during the hospital stage | from admission to discharge or death during reference hospitalization, assessed up to 90 days
Rehospitalization due to pneumonia, COVID-19, flu and other acute respiratory infections (ARV) | from discharge up to two years after reference hospitalization
  proportion of patients with rehospitalization due to pneumonia, COVID-19, flu and other acute respiratory infections (ARV)
Hospitalization due to cardiovascular disease (CVD) | from discharge up to two years after reference hospitalization
  proportion of patients with hospitalization due to cardiovascular disease
time to Flu and other ARV (except COVID-19) | from discharge up to two years after reference hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, MD, PhD, Study Chair — National Medical Research Center for Therapy and Preventive Medicine; Mikhail Loukianov, MD, PhD, Study Chair — National Medical Research Center for Therapy and Preventive Medicine; Andrey Pulin, MD, PhD, Study Chair — National Medical and Surgical Center named after N.I.Pirogov
Locations (2):
- Russia (2):
  - National Research Center for Preventive Medicine of the Ministry of Health, Moscow
  - National Medical and Surgical Center named after N.I.Pirogov of the Ministry of Health of Russian Federation, Moscow

REFERENCES:
- [Result] Drapkina O. M., Karpov O. E., Lukyanov M. M., Martsevich S. Yu., Pulin A. A., Kutishenko N. P., Akimkin V. G., Andreenko E. Yu., Voronina V. P., Dindikova V. A., Dmitrieva N. A., Zagrebelnyi A. V., Ler- man O. V., Makoveeva A. N., Okshina E. Yu., Kudryashov E. V., Klyashtorny V. G., Smirnov A. A., Fomina V. S. Prospective in-hospital registry of patients with suspected or documented COVID-19 infection and community acquired pneumonia (TARGET-VIP): characteristics of patients and assessment of in-hospital outcomes. Cardiovascular Therapy and Prevention. 2020;19(6):2727. (In Russ.) doi:10.15829/1728-8800-2020-2727
- [Result] Drapkina OM, Karpov OE, Loukyanov MM, Martsevich SYu, Pulin AA, Kutishenko NP, Akimkin VG, Andreenko EYu, Voronina VP, Dindikova VA, Dmitrieva NA, Zagrebelnyy AV, Lerman OV, Makoveeva AN, Okshina EYu, Kudryashov EV, Klyashtorniy VG, Smirnov AA, Fomina VS. Experience of creating and the first results of the prospective hospital registry of patients with suspected or confirmed coronavivirus infection (COVID-19) and community-acquired pneumonia (TARGET-VIP). The Russian Journal of Preventive Medicine. 2020;23(8):6- 13. (In Russ.). https://doi.org/10.17116/profmed2020230816
- [Result] Lukyanov M.M., Martsevich S.Yu., Pulin A.A., Kutishenko N.P., Andreenko E.Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Zagrebelny A.V., Makoveeva A.N., Lerman O.V., Okshina E.Yu., Sgibneva A. S., Smirnov A. A., Belova E. N., Klyashtorny V. G., Kudryashov E.V., Karpov O.E., Drapkina O.M. Dynamics of age characteristics and prevalence of concomitant cardiovascular and non-сardiovascular diseases in patients hospitalized with COVID-19 during epidemic wave: data from TARGET-VIP registry. Cardiovascular Therapy and Prevention. 2021;20(8):3106. (In Russ.) doi:10.15829/1728-8800-20213106
- [Result] : Martsevich S.Yu., Lukyanov M.M., Pulin A.A., Kutishenko N.P., Andreenko E.Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Zagrebelnyy A.V., Lerman O.V., Makoveeva A.N., Okshina E.Yu., Smirnov A.A., Kudryashov E.V., Budaeva I.V., Nikoshnova E.S., Karpov O.E., Drapkina O.M. Prehospital Period in Patients with COVID-19: Cardiovascular Comorbidity and Pharmacotherapy During the First Epidemic Wave (Hospital Registry Data). Rational Pharmacotherapy in Cardiology 2021;17(6):873-879. DOI:10.20996/1819-6446-2021-12-13
- [Result] Lukyanov M.M., Kutishenko N.P., Martsevich S.Yu., Pulin A.A., And - reenko E. Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Lerman O.V., Makove - eva A.N., Okshina E.Yu., Sgibneva A.S., Smirnov A.A., Belova E.N., Klyashtorny V.G.,Kudryashov E.V., Karpov O.E., Drapkina O.M. Long-term outcomes in patients after COVID-19: data from the TARGET-VIP registry. Russian Journal of Cardiology. 2022;27(3):4912. doi:10.15829/1560-4071-2022-4912
- [Result] Smirnov A.A., Loukianov M.M., Martsevich S.Yu., Pulin A.A., Kutishenko N.P., Andreenko E.Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Kudryavtseva M.M., Lerman O.V., Makoveeva A.N., Okshina E.Yu., Maltseva A.A., Belova E.N., Klyashtorniy V.G., Kudryashov E.V., Karpov O.E., Drapkina O.M. Clinical and Anamnestic Characteristics, Cardiovascular Pharmacotherapy and Long-term Outcomes in Multimorbid Patients after COVID-19. Rational Pharmacotherapy in Cardiology 2022;18(5):502-509. DOI:10.20996/1819-6446-2022-09-06
- [Result] Loukyanov MM, Andreenko EYu, Martsevich SYu, Kutishenko NP, Voronina VP, Dindikova VA, Dmitrieva NA, Kudryavtseva MM, Lerman OV, Makoveeva AN, Okshina EYu, Smirnov AA, Belova EN, Kudryashov EV, Litinskaya OA, Dzodzuashvili LR, Karpov OE, Pulin AA, Drapkina OM. Long-term follow-up of patients after COVID-19: adherence to SARS-CoV-2 vaccination and immune status. Profilakticheskaya Meditsina. 2022;25(12):88-95. (In Russ.). https://doi.org/10.17116/profmed20222512188
- [Result] Kutishenko N.P., Lukyanov M.M., Martsevich S.Yu., Pulin A.A., Andreenko E.Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Kudryavtseva M.M., Lerman O.V., Makoveeva A.N., Okshina E.Yu., Smirnov А.А., Belova E.N., Klyashtorny V.G., Kudryashov E.V., Karpov O.E., Drapkina O.M. Medical treatment of patients with cardiovascular diseases during the first year after hospitalization for COVID-19. Cardiovascular Therapy and Prevention. 2022;21(12):3467. (In Russ.) https://doi.org/10.15829/1728-8800-2022-3467
- [Result] Mareev Yu.V., Lukyanov M.M., Martsevich S.Yu., Pulin A.A., Kutishenko N.P., Andreenko E.Yu., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Makoveeva A.N., Lerman O.V., Okshina E.Yu., Smirnov A.A., Kudryavtseva M.M., Belova E.N., Klyashtorny V.G., Kudryashov E.V., Karpov O.E., Drapkina O.M. Detection rate and characteristics of heart failure, depending on the diagnostic criteria in COVID-19 survivors one year after hospitalization. Cardiovascular Therapy and Prevention. 2022;21(12):3437. (In Russ.) https://doi.org/10.15829/1728-8800-2022-3437
- [Result] Lukyanov M.M., Andreenko E. Yu., Martsevich S. Yu., Kutishenko N.P., Voronina V.P., Dindikova V.A., Dmitrieva N.A., Kudryavtseva M.M., Lerman O.V., Makoveeva A.N., Okshina E. Yu., Pulin A.A., Smirnov A.A., Klyashtorny V.G., Karpov O.E., Drapkina O.M. Two-year outcomes in patients after hospitalization for COVID-19: data from the TARGET-VIP registry. Cardiovascular Therapy and Prevention. 2023;22(10):3757. doi:10.15829/1728-8800-2023-3757
- [Result] Smirnov AA, Loukianov MM, Martsevich SYu, Kutishenko NP, Andreenko EYu, Voronina VP, Dindikova VA, Dmitrieva NA, Kudryavtseva MM, Lerman OV, Makoveeva AN, Okshina EYu, Smirnova MI, Pulin AA, Karpov OE, Drapkina OM. Long-term outcomes in patients with cardiovascular multimorbidity suffered from COVID-19: two-year observation. The Russian Journal of Preventive Medicine. 2023;26(12):58-64. (In Russ.). https://doi.org/10.17116/profmed20232612158